CLINICAL TRIAL: NCT00332722
Title: Effectiveness of Cervical Facet Joint Nerve Blocks: A Randomized, Prospective, Double-Blind Controlled Evaluation
Brief Title: Effectiveness of Cervical Facet Joint Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, C.E.O, Pain Management Center of Paducah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol4
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Results first posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1- without steroid (Active Comparator): Cervical Facet Joint Nerve block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin)
  Interventions: Procedure: Cervical facet joint nerve blocks
- Group 2 - with steroid (Active Comparator): Cervical Facet Joint nerve block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin) and 0.15 mg of non-particulate betamethasone)
  Interventions: Procedure: Cervical facet joint nerve blocks

INTERVENTIONS:
Procedure: Cervical facet joint nerve blocks

SUMMARY:
1. To demonstrate whether:

   i. Facet joint nerve blocks have therapeutic value beyond the duration of local anesthetic effect.

   ii. Adjuvant medications (Sarapin and Depo-Medrol) provide additional relief of cervical facet joint pain when used with facet joint nerve blocks.
2. To demonstrate whether or not there are clinically significant improvements in function of patients who receive cervical facet joint nerve block with or without Sarapin and Depo-Medrol (Group II) compared to patients randomized to Group I who receive only local anesthetic blocks.
3. To determine the adverse event profile in both groups.

ELIGIBILITY:
Inclusion Criteria:

Positive for facet joint pain with comparative local anesthetic blocks

Candidates are over 18 years of age

Subjects with a history of chronic, function limiting neck pain of at least six months in duration Subjects who are able to give voluntary, written informed consent to participate in this investigation Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the center for all the required post-operative follow-ups The subject has not had recent surgical procedures within the last three months.

Exclusion Criteria:

Negative or false-positive response to controlled comparative local anesthetic blocks

Narcotic use of greater than Hydrocodone 100 mg/day, Methadone 80 mg or Morphine 100 mg, or dose equivalent

Uncontrolled major Depression or uncontrolled psychiatric disorders

Uncontrolled or acute medical illnesses including coagulopathy, renal insufficiency, chronic liver dysfunction, progressive neurological deficit, urinary sphincter dysfunction, infection, increased intercranial pressure, pseudotumor cerebri, intercranial tumors, unstable angina, and severe chronic obstructive pulmonary disease.

Chronic severe conditions that could interfere with the interpretations of the outcome assessments for pain and bodily function

Women who are pregnant or lactating

Subjects who have participated in a clinical study with an investigational product within 30 days of enrollment

Patients with multiple complaints involving concomitant hip osteoarthritis, will not be amenable to study due to the overlap of pain complaints.

Inability to achieve appropriate positioning and inability to understand informed consent and protocol History of adverse reaction to local anesthetic or anti-inflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-09; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States

REFERENCES:
- [Result] Manchikanti L, Singh V, Falco FJ, Cash KA, Fellows B. Comparative outcomes of a 2-year follow-up of cervical medial branch blocks in management of chronic neck pain: a randomized, double-blind controlled trial. Pain Physician. 2010 Sep-Oct;13(5):437-50. PMID 20859313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive new patients presenting to interventional pain management practice with neck pain without suspected disc herniation or radiculitis.
Groups:
- Group 1 Without Steroids: Cervical Facet Joint nerve block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin)
- Group 2 With Steroids: Cervical Facet Joint nerve block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin) and 0.15 mg of non-particulate betamethasone)
Period: Overall Study
Arm/Group | Group 1 Without Steroids | Group 2 With Steroids
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1- Without Steroid | Group 2 - With Steroid | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (13.2) | 43 (14.1) | 44 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 48 | 89
  Male | 19 | 12 | 31
duration of pain [Mean (Standard Deviation); unit: months] | 120 (122) | 87 (104) | 103 (174)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS)
Description: Numeric Rating Scale (range 0-10) is represented as 0 for no pain and 10 for worst pain imaginable.
Time Frame: over 2 years
Population: A sample size of 60 patients for each group was chosen.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1 - Without Steroids: Cervical Facet Joint nerve block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin)
- Group 2 - With Steroids: Cervical Facet Joint nerve block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin) and 0.15 mg of non-particulate betamethasone)
Arm/Group | Group 1 - Without Steroids | Group 2 - With Steroids
Number analyzed (Participants) | 60 | 60
units on a scale
  Baseline | 8.2 (0.8) | 8.2 (1.1)
  2 years | 3.5 (1.1) | 3.2 (1.0)
Statistical Analysis 1: Comparison: Group 1 - Without Steroids vs Group 2 - With Steroids; Test type: Superiority or Other; p < 0.05, Paired t test

2. Secondary Outcome: Neck Disability Index (NDI)
Description: Neck Disability Index (range 0-50) is represented as 0-4 no disability, 5-14 mild disability, 15 - 24 moderate disability, 25 - 34 severe disability and >34 (35-50) complete disability.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - Without Steroids | Group 2 - With Steroids
Number analyzed (Participants) | 60 | 60
units on a scale
  Baseline | 25.4 (5.7) | 25.1 (5.0)
  24 months | 11.6 (5.2) | 11.0 (4.7)
Statistical Analysis 1: Comparison: Group 1 - Without Steroids vs Group 2 - With Steroids; Test type: Superiority or Other; p < 0.05, Paired t test

ADVERSE EVENTS:
Time Frame: 24 months
Description: Infection, Nerve root or Spinal cord trauma
Arm/Group | Group 1- Without Steroid | Group 2 - With Steroid
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- Without Steroid (N=60) | Group 2 - With Steroid (N=60)
Infection (Infections and infestations) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study limitations include the lack of a placebo group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No